CLINICAL TRIAL: NCT06159855
Title: The Effect of Bowel Preparation Training Given to Patients Planned to Undergo Colonoscopy and the Monitoring Carried Out by the Nurse on Anxiety, Compliance With Bowel Preparation and Bowel Cleansing
Brief Title: The Effect of Bowel Preparation Training Given to Patients Undergoing Colonoscopy
Acronym: training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BBUYUKKILIC
Record Dates: First submitted 2023-11-08; First posted 2023-12-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-08

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Group: Data Collection (Other): 1. PRE-TEST
     a) Who is decided to have a colonoscopy, using the Patient Information Survey, Procedure Compliance Survey and Beck Anxiety Scale.
  2. ROUTINE APPLICATION
     1. Patients who are planned to undergo colonoscopy and are included in the control group will be trained according to the bowel preparation protocol routinely applied by the clinical nurse.
     2. The Procedure Compliance Survey, which is routinely used as a clinical procedure, is given to the patient/patient's relative after the training of the clinical nurse.
  3. FINAL TEST
     1. Immediately after the procedure, data will be collected again with the Patient Information Survey, Procedure Compliance Survey and Beck Anxiety Scale.
     2. After the procedure, the cleanliness of the intestines will be evaluated by the physician with the Ottawa Bowel Preparation Scale.
     3. The control group will be given training and a booklet after all data collection is completed.
  Interventions: Other: Intervention group: nurse-led education for bowel preparation of colonoscopy

INTERVENTIONS:
Other: Intervention group: nurse-led education for bowel preparation of colonoscopy — 1. PRE-TEST
     a) Patients will be evaluated using the Patient Information Survey, Procedure Compliance Survey and Beck Anxiety Scale.
  2. INTERVENTION
     1. Patients will be given face-to-face training in the clinic training room of the unit.
     2. After face-to-face training is given, an educational brochure will be given to the patient.
     3. If the patient is constipated, the bowel preparation diet is requested to be started 5 days in advance. If the patient is not constipated, the bowel preparation diet is started 3 days in advance.
     4. After the intervention group is given bowel preparation training, reminders about colonoscopy will be made via instant messaging 3 to 5 days before the day of the colonoscopy.
  3. LAST TEST
     1. Data will be collected again using the Patient Information Survey, Procedure Compliance Survey and Beck Anxiety Scale.
     2. The cleanliness of the intestines will be evaluated by the physician using the Ottawa Bowel Preparation Scale.

SUMMARY:
This study was planned to examine the effect of bowel preparation training and monitoring given to patients planned to undergo colonoscopy on the level of anxiety, compliance with bowel preparation and bowel cleansing. The research sample was collected at the Sultan II. University of Health Sciences affiliated to the Istanbul Provincial Health Directorate between December 2022 and August 2023. 34 intervention and 34 control groups will be randomly selected from outpatients who apply to the Colonoscopy Unit of Abdülhamid Han Training and Research Hospital and meet the inclusion criteria.

In this study, it is aimed to increase the effect of bowel preparation training, supported by nurses in the clinic and via instant messaging/calling or communication application, on patients' anxiety level, level of compliance with bowel preparation, and bowel cleansing in patients scheduled for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy is planned
* Understands Turkish, can read and write,
* Patients who volunteer to participate in the research.

Exclusion Criteria:

* Patients who do not attend planned training and do not receive telephone counseling

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Survey | baseline, pre-intervention (pre-colonoscopy procedure)
  It includes data about the personal characteristics
Beck Anxiety Inventory | pre-intervention (pre colonoscopy procedure)
  It measures the level of anxiety before colonoscopy prosedure
Procedure Compliance Survey | immediately post-intervention (post colonoscopy procedure)
  It measures the level of compliance to interventions after colonoscopy prosedure
Ottawa Bowel Preparation Scale | immediately post-intervention (post colonoscopy procedure)
  It is used to assess a patient's bowel preparation for colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science, Istanbul, Uskudar, Turkey (Türkiye)

REFERENCES:
- [Background] Wang C, Xie XL, Hou DC, Sun C, He WY. Effect of WeChat Messaging on Improving the Quality of Bowel Preparation for Outpatient Colonoscopy: A Randomized Controlled Study. Gastroenterol Nurs. 2022 Mar-Apr 01;45(2):120-126. doi: 10.1097/SGA.0000000000000625. PMID 35283439
- [Background] Lee E, Shafer LA, Walker JR, Waldman C, Michaud V, Yang C, Bernstein CN, Hathout L, Park J, Sisler J, Wittmeier K, Restall G, Singh H. Information experiences, needs, and preferences of colonoscopy patients: A pre-colonoscopy survey. Medicine (Baltimore). 2019 May;98(20):e15738. doi: 10.1097/MD.0000000000015738. PMID 31096537
- [Background] Xu F, Lu S, Dong L, He Y, Li H, Tang J. Educational Video on the WeChat Platform Can Effectively Improve the Quality of Bowel Preparation: A Prospective, Randomized, Controlled Study. Gastroenterol Nurs. 2021 Jan-Feb 01;44(1):47-51. doi: 10.1097/SGA.0000000000000528. PMID 33351522
- [Background] Mahmud N, Asch DA, Sung J, Reitz C, Coniglio MS, McDonald C, Bernard D, Mehta SJ. Effect of Text Messaging on Bowel Preparation and Appointment Attendance for Outpatient Colonoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2034553. doi: 10.1001/jamanetworkopen.2020.34553. PMID 33492374
- [Background] Wang SL, Wang Q, Yao J, Zhao SB, Wang LS, Li ZS, Bai Y. Effect of WeChat and short message service on bowel preparation: an endoscopist-blinded, randomized controlled trial. Eur J Gastroenterol Hepatol. 2019 Feb;31(2):170-177. doi: 10.1097/MEG.0000000000001303. PMID 30418256